CLINICAL TRIAL: NCT02025595
Title: The Role of Central Reward and Satiety Centers in the Etiology of Obesity: Genetic and Environmental Influences
Brief Title: Obesity and Brain: Genes and Environment
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, RG IJzerman, MD PhD FRCPE, Professor of Internal Medicine, Chair of Diabetology, Director of Diabetes Center VUmc, Amsterdam UMC, location VUmc
Other Study IDs: DC2013ObesiBrain001; NL 44735.029.13 (Other: The Central Committee on Research Involving Human Subjects (CCMO)); 91613082 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2013-12-13; First posted 2014-01-01 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: Brain; Genes; Environment; Etiology; Reward; Satiety Response; Central Nervous System; Magnetic Resonance Imaging; Twins, Monozygotic; Overweight; Obesity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Monozygotic twin pairs: 15 monozygotic twin pairs discordant for obesity
- Genetic predisposition for obesity: 15 obese and 15 non-obese individuals with a high genotype obesity risk score and 15 obese and 15 non-obese individuals with a low genotype obesity risk score. Genotype obesity risk score will be based on genome wide association single-nucleotide polymorphisms (SNP's) associated with obesity.

SUMMARY:
The aim of this study is to investigate the effects of genetic and environmental risk factors on central nervous system (CNS) reward and satiety circuits in the etiology of obesity. The investigators will also investigate to what extent the alterations in CNS reward and satiety circuits are a cause or a consequence of the development of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Male or female
* Stable bodyweight (<5% reported weight change during previous 3 months)
* Women: regular menstruation cycle (to exclude possible menstruation cycle effects)
* Normal fasting blood glucose

Exclusion Criteria:

* Left handedness
* Known diabetes or abnormal fasting blood glucose
* Serious heart, pulmonary, hepatic or renal disease, malignant or hematological disease
* Metabolic disorders (uncontrolled adrenal/thyroid disease)
* Women: irregular menstruation cycle
* Neurological or psychiatric illness
* Pregnancy or breast feeding
* Alcohol abuse
* Nicotine abuse
* Claustrophobia or metal implants
* Visual disability
* Participation in another study
* Inability to understand the protocol or to give informed consent
* Current/chronic use of following medication: antihyperglycemic agents, glucocorticoids, centrally acting drugs, cytostatics, immune suppressants, potentially addictive medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Netherlands Twin Registry (NTR). All subjects are voluntary participants and have received surveys on lifestyle and health every 2 years. In addition, genome wide data are available in a large number of these individuals.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The difference in neuronal activity in CNS reward and satiety circuits as represented by BOLD functional magnetic resonance imaging (fMRI) signal change from baseline (%) in response to food-related stimuli within obesity discordant MZ twin pairs. | Baseline (one measurement)
The difference in neuronal activity in CNS reward and satiety circuits as represented by BOLD fMRI signal change from baseline (%) in response to food-related stimuli between individuals at high verses low genetic obesity risk. | Baseline (one measurement)
The difference in neuronal activity in CNS reward and satiety circuits as represented by BOLD fMRI signal change from baseline (%) in response to food-related stimuli between lean and obese subjects with either high or low genetic obesity risk. | Baseline (one measurement)

SECONDARY OUTCOMES:
The difference within obesity-discordant monozygotic (MZ) twin pairs regarding dietary intake | Baseline (one measurement)
  Dietary intake will be measured as quantitative (kcal/day) and qualitative (energy density (kcal/kg) and macronutrient composition (%)) dietary intake using A) a choice lunch buffet on the visit day and B) the 24 hours recall method on two week days and one weekend day at home.
The difference within obesity-discordant monozygotic (MZ) twin pairs regarding physical activity level | Baseline (one measurement)
  Physical activity level will be measured as metabolic equivalent of task (METs)-hours per week using seven-day ActiGraph triaxial accelerometry at home.
The difference within obesity-discordant monozygotic (MZ) twin pairs regarding basal metabolic rate | Baseline (one measurement)
  Basal metabolic rate will be measured in kcal/day using oxygen consumption and carbon dioxide production measured by indirect calorimetry using a ventilated hood system.
The difference within obesity-discordant monozygotic (MZ) twin pairs regarding fasting circulating biomarker levels | Baseline (one measurement)
  Fasting circulating biomarker levels (glucose (mmol/l), HbA1c (mmol/mol), insulin (pmol/l), C-peptide (nmol/l), glucagon (pmol/l), triglycerides (mmol/l), HDL-cholesterol (mmol/l) and LDL-cholesterol (mmol/l)) will be measured in a fasting blood sample.
The difference within obesity-discordant monozygotic (MZ) twin pairs regarding autonomic nervous system balance | Baseline (one measurement)
  Autonomic nervous system balance will be assessment based on measurements of A) heart rate variability (HRV; calculated as root mean square of successive R-R interval differences (RMSSD) in ms2); B) respiratory rate (RR; breaths/min) and C) respiratory sinus arrhythmia (RSA; ms) in resting conditions and in response to a mental arithmetic task using an electro- and impedance cardiogram.
The difference between individuals at high versus those at low genetic obesity risk regarding dietary intake | Baseline (one measurement)
  Dietary intake will be measured as quantitative (kcal/day) and qualitative (energy density (kcal/kg) and macronutrient composition (%)) dietary intake using A) a choice lunch buffet on the visit day and B) the 24 hours recall method on two week days and one weekend day at home.
The difference between individuals at high versus those at low genetic obesity risk regarding physical activity level | Baseline (one measurement)
  Physical activity level will be measured as metabolic equivalent of task (METs)-hours per week using seven-day ActiGraph triaxial accelerometry at home.
The difference between individuals at high versus those at low genetic obesity risk regarding basal metabolic rate | Baseline (one measurement)
  Basal metabolic rate will be measured in kcal/day using oxygen consumption and carbon dioxide production measured by indirect calorimetry using a ventilated hood system.
The difference between individuals at high versus those at low genetic obesity risk regarding fasting circulating biomarker levels | Baseline (one measurement)
  Fasting circulating biomarker levels (glucose (mmol/l), HbA1c (mmol/mol), insulin (pmol/l), C-peptide (nmol/l), glucagon (pmol/l), triglycerides (mmol/l), HDL-cholesterol (mmol/l) and LDL-cholesterol (mmol/l)) will be measured in a fasting blood sample.
The difference between individuals at high versus those at low genetic obesity risk regarding autonomic nervous system balance | Baseline (one measurement)
  Autonomic nervous system balance will be assessment based on measurements of A) heart rate variability (HRV; calculated as root mean square of successive R-R interval differences (RMSSD) in ms2); B) respiratory rate (RR; breaths/min) and C) respiratory sinus arrhythmia (RSA; ms) in resting conditions and in response to a mental arithmetic task using an electro- and impedance cardiogram.

OTHER OUTCOMES:
The difference within obesity-discordant monozygotic (MZ) twin pairs regarding gut microbiota composition | Baseline (one measurement)
  Gut microbiota composition (ratio between various gut microbiota species) will be assessed by identifying microbial phylotypes in a feces sample using 16S ribosomal RNA molecule-based approaches of diagnostic analysis. Function of gut microbiota will be investigated using metaproteomics analysis techniques that include mass-spectroscopy methodologies.
  Please note: this outcome measure is conditional to available budget.
The difference within obesity-discordant monozygotic (MZ) twin pairs regarding epigenetic changes | Baseline (one measurement)
  Epigenetic changes will be assessed by measuring global DNA methylation (%) and locus specific DNA methylation (%) in regions of selected loci using a mass spectrometry-based method. Loci will be selected on the basis of their previously shown features of epigenetic regulation and their involvement in cardiovascular and metabolic disease.
  Please note: this outcome measure is conditional to available budget.
The difference between individuals at high versus those at low genetic obesity risk regarding gut microbiota composition | Baseline (one measurement)
  Gut microbiota composition (ratio between various gut microbiota species) will be assessed by identifying microbial phylotypes in a feces sample using 16S ribosomal RNA molecule-based approaches of diagnostic analysis. Function of gut microbiota will be investigated using metaproteomics analysis techniques that include mass-spectroscopy methodologies.
  Please note: this outcome measure is conditional to available budget.
The difference between individuals at high versus those at low genetic obesity risk regarding epigenetic changes | Baseline (one measurement)
  Epigenetic changes will be assessed by measuring global DNA methylation (%) and locus specific DNA methylation (%) in regions of selected loci using a mass spectrometry-based method. Loci will be selected on the basis of their previously shown features of epigenetic regulation and their involvement in cardiovascular and metabolic disease.
  Please note: this outcome measure is conditional to available budget.

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Doornweerd S, De Geus EJ, Barkhof F, Van Bloemendaal L, Boomsma DI, Van Dongen J, Drent ML, Willemsen G, Veltman DJ, IJzerman RG. Brain reward responses to food stimuli among female monozygotic twins discordant for BMI. Brain Imaging Behav. 2018 Jun;12(3):718-727. doi: 10.1007/s11682-017-9711-1. PMID 28597337
- [Derived] Doornweerd S, IJzerman RG, van der Eijk L, Neter JE, van Dongen J, van der Ploeg HP, de Geus EJ. Physical activity and dietary intake in BMI discordant identical twins. Obesity (Silver Spring). 2016 Jun;24(6):1349-55. doi: 10.1002/oby.21475. Epub 2016 Apr 23. PMID 27106364